CLINICAL TRIAL: NCT04118790
Title: New Clinical Magnetic Resonance Technologies for Capturing Brain Microstructure Alterations in Patients With Minor Stroke or Transient Ischemic Attack
Brief Title: Microstructure Imaging in Stroke Patients
Status: Recruiting | Type: Observational
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Tim Dyrby, Senior Researcher, Danish Research Centre for Magnetic Resonance
Other Study IDs: TRABIT13
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Fatigue; Stroke, Acute; Transient Ischemic Attack
Keywords: Fatigue; minor stroke; TIA; Diffusion; MRI; Quantitative; Sequence; Microstructure; Axon; Myelin; Degeneration
MeSH Terms: conditions — Fatigue; Stroke; Ischemic Attack, Transient | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Minor Stroke patients: * Clinical Assessment
  * MRI scan session
  Interventions: Other: Clinical Assessment; Procedure: MRI scan
- TIA patients: * Clinical Assessment
  * MRI scan session
  Interventions: Other: Clinical Assessment; Procedure: MRI scan
- Healthy Controls: * MRI scan session
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Other: Clinical Assessment — 1. Medical history and details of the vascular incident will be collected from the patient and the medical journal. (Duration: 1hr)
  2. Neuropsychological measures collected using test measures and questionaries (duration approx 45-60 min).
  Groups: Minor Stroke patients; TIA patients
Procedure: MRI scan — 1. MRI scan session, which includes Structural, Quantitative, Functional and Diffusion MRI sequences. (maximum duration: 90 min).

SUMMARY:
The purpose of this study is to establish a methodological framework based on existing advanced neuroimaging technologies as a new clinical neuroimaging tool for assessment of possible affected brain connections in stroke and TIA patients. Thus, providing new insights into microstructural changes that may underline why those patients experience deficits like fatigue.

DETAILED DESCRIPTION:
Background:

Stroke and transient ischemic attack (TIA) patients are often burdened by fatigue and reduced attention span subacutely. The frequency of post-stroke fatigue is estimated to occur in 29-77% of all patients, with the highest burden often reported at 3 months post-stroke. The micro-sized structures that form the brain connection, i.e. White Matter (WM), the low blood flow, and the little collateral blood supply make the WM highly susceptible to ischemic injuries. In the case of stroke or TIA in WM, the surrounding microstructures of the are affected start losing vital nutrients, i.e. oxygen and glucose, which initiate a cascade of cellular dysfunction due to excitotoxicity. As a result, several microstructures deteriorate and degenerate, leading to neuronal damage and reduction of signal conduction. Diagnosis of stroke and TIA relies on clinical findings and imaging, where MRI has become the chosen imaging modality due to the sensitivity to detect brain lesions. However, at the later sub-acute phases of stroke and TIA, the standard clinical MRI sequences lack specificity to map microstructural degeneration/regeneration of the brain connections that project through or nearby the ischemic area. In recent years, new technologies for structural quantitative MRI have emerged that are sensitive to different microstructural features and their anisotropy organization i.e. demyelination and axonal sizes and densities. Using these new MRI methods has the potential to disentangle some of the pathological processes underlying minor stroke phases in a more quantitative way. Previously, a similar MRI study of future directions of clinical MRI technologies was applied to the Multiple Sclerosis disease (MS). The MS disease follows some of the systemic pathological degeneration effects as in minor stroke i.e. axonal degeneration and de-/remyelination. The preliminary results of that study strongly suggest e.g. that the newly introduced MRI modality improves diagnostic value by better correlation with clinical assessment. Furthermore, the combination of MRI modalities provides new insight into pathology only seen in histology.

Objectives:

1. To investigate whether new MRI methods can detect the impact of microstructure ischemic changes along brain connections e.g. neuronal degeneration.
2. To test the hypothesis that a combination of unique structural MRI measures will synergistically provide patterns of altered brain structure that give rise to excessive fatigue in patients with minor stroke or TIA.
3. To evaluate the capability of the new quantitative MRI methods to objectively assess the presence and severity of fatigue by pinpointing the relevant structural brain alterations that contribute to fatigue.

Hypothesis:

The central hypothesis of the study is that a combination of unique MRI measures will synergistically provide a stronger tool to describe the fatigue and cognitive deficits after stroke and TIA in order to predict the functional deficits in minor stroke and TIA. The assumption is that both Wallerian degeneration and demyelination are expected to affect the anisotropy of microstructural measures along the brain network, as they are inferred from diffusion processes on a micrometer length scale.

Methods:

* Participants: 90 participants are expected to be enrolled in this study. The participants are divided by the case-control method to form in total a 3 class group: 30 minor stroke patients, 30 TIA patients, and 30 healthy age- and sex-matched subjects for the control group.
* MRI sequences: Structural MRI (FLAIR, T1-W, T2*, and Magnetization Transfer), Quantitative MRI (Multiparametric mapping), and Diffusion-weighted imaging ( Diffusion Tensor Imaging, Tractography, Neurite Orientation Dispersion and Density Imaging (NODDI) model, and Microscopic Fractional Anisotropy).
* Neuropsychological measures: Fatigue score, estimated by Multidimensional Fatigue Inventory; Depression score, estimated by Major Depression Inventory; Fatigue Scale for Motor and Cognitive Functions; Repeatable Battery for the Assessment of Neuropsychological status; Wechsler Memory Scale-III; Verbal fluency tasks measuring semantic fluency; and Trail making test A and B.

Experimental Design:

* Part 1. Clinical and Cognitive assessment The clinical and cognitive assessments will be carried out at the Department of Neurology at Bispebjerg Hospital. The evaluation of cognitive assessment will be done through a series of tasks and questionnaires, which determine if the patient is eligible for the study.
* Part 2. MRI session The second part will take place within 3 weeks after the clinical assessment of the patients and consist of only 1 scan session. Healthy controls subjects will be included only for this second part with the aim to generate a reference frame of the imaging results on how the normal brain appears. The scan session has a maximum duration of 90 minutes.

Ethical Considerations:

All patients are handled according to best clinical practice and in accordance with Danish and European guidelines. There is no known risk related to MRI in persons with no magnetic metal in the body (e.g. a pacemaker); this is excluded by using a specific questionnaire to screen subjects prior to MRI. The confined space and the noise of the MRI-scanner may cause anxiety in some; therefore, all subjects will be provided with earplugs, and they must not suffer from claustrophobia. The investigators are not responsible for failure to find existing pathology in the MRI scans. However, on occasion the investigator may notice an incidental finding on an MRI scan that seems abnormal, a radiologist will be consulted as to whether the finding merits further investigation, in which case the investigator will contact the participant and/or the primary care physician of the participant to inform the finding. The decision as to whether to proceed with further examination or treatment lies solely with the participant and, if applicable, with the physician of the participant.

Economy:

The project has received funding from the European Union's Horizon 2020 research and innovation program under the Marie Skłodowska-Curie grant agreement No. 765148, European Innovative Training Network (ITN) program entitled TRABIT - "Translational Brain Imaging Training Network".

Importance or relevant to the study:

If the hypotheses of the study are confirmed, MRI-based fatigue imaging will provide an important addition to the clinical assessment based on clinical scores of the subjective perception of fatigue. Such MRI-based methods would pave the way for quantitative measurement of disabling fatigue and thus foster the development and assessment of individualized therapies.

ELIGIBILITY:
Patient Inclusion Criteria:

* Stroke or TIA (ABCD2>4 and/or acute Diffusion-Weighted Image (DWI) lesion).
* Modified Rankin Scale <=2.
* As perceived by the investigator, have the ability to comply with all requirements of the study protocol.
* Have the ability to understand and sign the Informed Consents Form.
* Multidimensional Fatigue Inventory score >= 12 on general fatigue.

Patient Exclusion Criteria:

* The DRCMR´s general exclusion criteria for MRI research.
* Pregnancy or lactation; human chorionic gonadotropin (hCG) urine test is offered for women < 55 years.
* Major medical illness (for instance: anemia, diabetes mellitus, thyroid disorders, cardiovascular disease, electrolyte imbalance, etc.)
* Treated with ritalin or modafinil.
* Known uncontrolled severe malignancy.
* Known drug or alcohol addiction.
* Tiredness due to pharmaceutical side effects, as identified by the Investigator.
* Max body weight of 130 kg.
* Persons who do not wish to be informed about abnormal findings as part of the investigations.

Healthy Controls Exclusion Criteria:

* The DRCMR´s general exclusion criteria for MRI research.
* Pregnancy or lactation; urin hCG test is offered for women < 55 years.
* Major medical illness (for instance: anemia, diabetes mellitus, thyroid disorders, cardiovascular disease, electrolyte imbalance, etc.)
* Anamnestic infection (cystitis, influenza, pneumonia, etc) the last 3 weeks.
* Known malignancy.
* Known drug or alcohol addiction.
* Tiredness due to pharmaceutical side effects.
* Max body weight of 130 kg.
* Persons who do not wish to be informed about abnormal findings as part of the investigations.

Healthy Controls Inclusion Criteria:

* Healthy
* Age- and sex-matched to patient groups.
* As perceived by the investigator, have the ability to comply with all requirements of the study protocol.
* Have the ability to understand and sign the Informed Consents Form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is in total 90 participants, from which, 3 groups are divided: 30 minor Stroke patients, 30 TIA patients, and 30 healthy controls.
  * The 2 groups of patients, minor Stroke and TIA, will be recruited from Department of Neurology, Bispebjerg Hospital.
  * The healthy age- and sex-matched individuals for the control group will be recruited from the general population.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Microstructural changes in the brain network, and its correlate with functional deficits in patients with minor stroke or TIA. | MRI data collected within 3 weeks after the clinical assessment
  The study assumes that minor stroke or TIA leads to both axonal Wallerian degeneration and demyelination. These pathological changes in the white matter brain network can be captured with a new microstructural anisotropy MRI measure related to cell density, shapes, and a measure of myelination. Therefore, a new microstructural fractional anisotropy measure is expected to be more sensitive to pathology than traditional estimations using the diffusion tensor models, such as diffusion tensor imaging (DTI). Moreover, the structural MRI measures are expected to correlate with clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Tim B. Dyrby, Professor, Principal Investigator — Danish Research Centre for Magnetic Resonance
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen, København NV
  - Danish Research Centre for Magnetic Resonance, Copenhagen

IPD SHARING:
Plan to Share IPD: No